CLINICAL TRIAL: NCT05932368
Title: Investigation of Early Change and Relationship Between Respiratory Functions, Respiratory Muscle Strength and Functional Capacities of Patients Undergoing Open Heart Surgery
Brief Title: Early Evaluation After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Yasemin Şahbaz, Lecturer, University of Beykent
Other Study IDs: UBeykent-4
Record Dates: First submitted 2023-06-20; First posted 2023-07-06 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Open Heart Surgery
Keywords: open heart surgery; respiratory functions; cardiac surgery; respiratory muscle strength; functional capacity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing open heart surgery: Patients who underwent open heart surgery at Istanbul University, Istanbul Medical Faculty, Department of Cardiovascular Surgery between 2018 and 2022, and whose data required for the study are complete in their discharge file.
  The inclusion criteria of the files were: the patient was between the ages of 25-70, had undergone open heart surgery, was included in a phase 1 cardiac rehabilitation program, and had a preoperative ejection fraction of over 40%. Files of patients who do not meet the inclusion criteria and do not give the necessary permission to use their data will not be included in the study.
  Interventions: Other: evaluation

INTERVENTIONS:
Other: evaluation — examining files and taking records

SUMMARY:
The aim of this study is to examine the changes in respiratory function, respiratory muscle strength and functional capacity markers and the relationship between them in patients who have undergone open heart surgery and are at the discharge stage.

Method: Preoperative and postoperative evaluation results of 34 patients at discharge will be examined. Evaluations in the file; demographic data, respiratory functions; It will include spirometric measurements and intraoral pressure measurements and functional capacity measurement results.

SPSS version 25 will be used in data analysis. The distribution of the participants according to their gender among the groups, presence of chronic diseases, regular drug use, smoking, alcohol use, regular exercise habits will be evaluated with the "chi-square" test. The conformity of the data to the normal distribution will be tested with the Shaphiro-Wilk Test.

The difference between before and after the operation will be evaluated with the Paired Sample T Test. Pearson Correlation Test was performed for the relationship between independent variables and the significance level will be accepted as p<0.05.

DETAILED DESCRIPTION:
The patient data analyzed for this retrospective study will be selected from the files of patients who underwent open heart surgery at Istanbul University, Istanbul Medical Faculty, Department of Cardiovascular Surgery and whose data required for the study were complete in their discharge file. Patient data between 2018 and 2022 will be reviewed and patients who consented to use their data for the study will be included in the study. Evaluation data of the patients before the operation and at the discharge stage after the operation will be drawn from the patient files. The study will be prepared in accordance with the Helsinki Declaration Criteria. Before starting the study, ethics committee approval was obtained from Istanbul University Istanbul Medical Faculty Clinical Research Ethics Committee (permission no: 1208327; date: 15/09/2022). All patients were informed verbally/written about the study and their written consents will be obtained.

The inclusion criteria of the files in the study will be determined as the patient's age between 25-70 years, having undergone open heart surgery, being included in a phase 1 cardiac rehabilitation program, and having an ejection fraction above 40% before the operation. Files of patients who do not meet the inclusion criteria and do not give the necessary permission to use their data will not be included in the study. Spirometric Measurements FVC, FEVı, FEVı%, PEF, FEF25-75 and MVV values, which were evaluated according to the ATS/ERS (American Thoracic Society/European Respiratory Society) criteria, where the highest results were recorded as a result of the measurements repeated 3 times in the PFT test, will be drawn from the patient files.

Intraoral Pressure Measurement Maximum inspiratory pressure (MIP), maximum expiratory pressure (MEP) values evaluated according to ATS/ERS criteria, where the highest results are recorded as a result of measurements repeated 3 times in the respiratory muscle strength test, will be drawn from the patient files. While interpreting the results, the normal values of inspiratory and expiratory muscle strength determined by age and gender will be taken and the percentage of the expected value will be used.

Functional Capacity 6-minute walk test (6MWT) Information about the test, which is applied in a 30-meter (m) long hospital corridor and the 6-minute walking distance of the patients is recorded, will be drawn from the patient file.

ELIGIBILITY:
Inclusion Criteria:

* The patient is between the ages of 25-70
* Having had open heart surgery
* Being enrolled in a phase 1 cardiac rehabilitation program
* Preoperative ejection fraction above 40%

Exclusion Criteria:

* Not meeting the inclusion criteria
* Who do not give the necessary permission to use their data

Ages: 25 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent open heart surgery at Istanbul University, Istanbul Faculty of Medicine, Department of Cardiovascular Surgery, and whose data required for the study are complete in their discharge file, will be selected from among the files. Patient data from 2018 to 2022 will be reviewed, and patients who have consented to use their data for the study will be included in the study. Evaluation data of the patients before the operation and at the discharge stage after the operation will be drawn from the patient files.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Spirometric Measurements-Forced vital capacity (FVC) | through study completion, an average of 1 months]
  FVC value, which was evaluated according to the ATS/ERS (American Thoracic Society/European Respiratory Society) criteria, where the highest results were recorded as a result of the measurements repeated 3 times in the PFT test, will be drawn from the patient files.
Spirometric Measurements-Forced expiratory volume (FEV1) | through study completion, an average of 1 months]
  Forced expiratory volume (FEV1) calculates the amount of air that a person can force out of their lungs in 1 second.
  FEV1 value, which was evaluated according to the ATS/ERS (American Thoracic Society/European Respiratory Society) criteria, where the highest results were recorded as a result of the measurements repeated 3 times in the PFT test, will be drawn from the patient files.
Spirometric Measurements-FEF25-75 | through study completion, an average of 1 months]
  FEF25-75 is the most sensitive measure of airflow in peripheral airways where primary airflow obstruction originates,7 and it is reduced in early bronchial impairment, which is associated with small airway disease.
  FEF25-75 value, which was evaluated according to the ATS/ERS (American Thoracic Society/European Respiratory Society) criteria, where the highest results were recorded as a result of the measurements repeated 3 times in the PFT test, will be drawn from the patient files.
Spirometric Measurements-MVV | through study completion, an average of 1 months]
  Formerly referred to as maximum breathing capacity, maximum voluntary ventilation (MVV) is a pulmonary function test (PFT) that measures the maximum amount of air a person can inhale and then exhale with voluntary effort
  MVV value, which was evaluated according to the ATS/ERS (American Thoracic Society/European Respiratory Society) criteria, where the highest results were recorded as a result of the measurements repeated 3 times in the PFT test, will be drawn from the patient files.
Spirometric Measurements--Peak Expiratory Flow (PEF) | through study completion, an average of 1 months]
  PEF value, which was evaluated according to the ATS/ERS (American Thoracic Society/European Respiratory Society) criteria, where the highest results were recorded as a result of the measurements repeated 3 times in the PFT test, will be drawn from the patient files.
Intraoral Pressure Measurement-MIP | through study completion, an average of 1 months]
  Maximum inspiratory pressure (MIP) value evaluated according to ATS/ERS criteria, where the highest results are recorded as a result of measurements repeated 3 times in the respiratory muscle strength test, will be drawn from the patient files. While interpreting the results, the normal values of inspiratory determined by age and gender were taken and the percentage of the expected value will be used.
Intraoral Pressure Measurement-MEP | through study completion, an average of 1 months]
  Maximum expiratory pressure (MEP) value evaluated according to ATS/ERS criteria, where the highest results are recorded as a result of measurements repeated 3 times in the respiratory muscle strength test, will be drawn from the patient files. While interpreting the results, the normal values of expiratory muscle strength determined by age and gender were taken and the percentage of the expected value will be used.

SECONDARY OUTCOMES:
Functional Capacity | through study completion, an average of 1 months]
  6-minute walk test (6MWT) Information about the test, which is applied in a 30-meter (m) long hospital corridor and the 6-minute walking distance of the patients is recorded, will be drawn from the patient file (ATS, 2016).

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. İpek Yeldan, Study Chair — Istanbul University - Cerrahpasa; Yasemin ŞAHBAZ, Principal Investigator — İstanbul Beykent Üniversitesi; Dr. Doğan Yetüt, Study Chair — Hakkari State Hospital, Cardiovascular Surgery, Hakkari; Pt. Tülin Özalhas, Study Chair — Istanbul University, Istanbul Faculty of Medicine, Department of Cardiovascular Surgery, Istanbul; Prof. Dr. İbrahim Ufuk Alpagut, Study Chair — Istanbul University, Istanbul Faculty of Medicine, Department of Cardiovascular Surgery, Istanbul
Locations (1):
- Beykent University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Miller MR, Crapo R, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. General considerations for lung function testing. Eur Respir J. 2005 Jul;26(1):153-61. doi: 10.1183/09031936.05.00034505. No abstract available. PMID 15994402
- [Result] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Result] Enright PL, Kronmal RA, Manolio TA, Schenker MB, Hyatt RE. Respiratory muscle strength in the elderly. Correlates and reference values. Cardiovascular Health Study Research Group. Am J Respir Crit Care Med. 1994 Feb;149(2 Pt 1):430-8. doi: 10.1164/ajrccm.149.2.8306041.